CLINICAL TRIAL: NCT06491485
Title: Magnesium Sulfate Versus Sodium Bicarbonate as Adjuvants to Lidocaine 1% by Intraperitoneal Instillation for Postoperative Analgesics in Laparoscopic Gynecological Surgeries
Brief Title: Postoperative Analgesia in Laparoscopic Gynecological Surgeries
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Hamza Abdelrady Abdelmalek, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Post laparoscopy analgesia
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain
Keywords: Laparoscopic gynecological surgeries
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Magnesium Sulfate; Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group M (Magnesium sulfate) (Experimental): a total volume 200 ml normal saline 0.9% at a temperature of 37°c including 3mg/kg of 1% lidocaine with magnesium sulfate 50 mg/kg (maximum 2g) will be sprayed by the surgeon through the laparoscopic port to wash the incisions and anastomosis.
  Interventions: Drug: Group M (lidocaine with Magnesium sulfate)
- Group B (Sodium bicarbonate) (Experimental): a total volume 200 ml normal saline 0.9% at a temperature of 37°c including 3mg/kg of 1% lidocaine with 50 ml 4.2% sodium bicarbonate will be sprayed by the surgeon through the laparoscopic port to wash the incisions and anastomosis.
  Interventions: Drug: Group B (lidocaine with Sodium bicarbonate)
- Group C (Active Comparator): a total volume 200 ml normal saline 0.9% at a temperature of 37°c including 3mg/kg of 1% lidocaine will be sprayed by the surgeon through the laparoscopic port to wash the incisions and anastomosis.
  Interventions: Drug: Group C (lidocaine with saline)

INTERVENTIONS:
Drug: Group M (lidocaine with Magnesium sulfate) — a total volume 200 ml normal saline 0.9% at a temperature of 37°c including 3mg/kg of 1% lidocaine with magnesium sulfate 50 mg/kg (maximum 2g) will be sprayed by the surgeon through the laparoscopic port to wash the incisions and anastomosis.
  Arms: Group M (Magnesium sulfate)
Drug: Group B (lidocaine with Sodium bicarbonate) — a total volume 200 ml normal saline 0.9% at a temperature of 37°c including 3mg/kg of 1% lidocaine with 50 ml 4.2% sodium bicarbonate will be sprayed by the surgeon through the laparoscopic port to wash the incisions and anastomosis.
  Arms: Group B (Sodium bicarbonate)
Drug: Group C (lidocaine with saline) — a total volume 200 ml normal saline 0.9% at a temperature of 37°c including 3mg/kg of 1% lidocaine will be sprayed by the surgeon through the laparoscopic port to wash the incisions and anastomosis.
  Arms: Group C

SUMMARY:
The aim of this study is to compare intraperitoneal instillation of magnesium sulfate versus sodium bicarbonate as an adjuvant to lidocaine 1% , on reducing postoperative pain in laparoscopic gynecological surgeries.

DETAILED DESCRIPTION:
Patients undergoing laparoscopic surgery experience postoperative pain especially in the abdomen, lower back, and shoulders, Relieving postoperative pain, especially with certain types of analgesic agents, may reduce postoperative morbidity and mortality. It is also important to prevent adverse events such as myocardial infarction, cardiac arrhythmia, ileus, and poor wound healing and pulmonary complications. There is evidence that the main source of pain after laparoscopic surgeries is the peritoneum . Due to CO2 insufflation constitutes the commonest means of creating the pneumoperitoneum. Co2pneumoperitoneum is known to cause systemic acidosis. Which is responsible for damaging of the mesothelial lining of the peritoneum and consequent peritoneal irritation . Moreover, the phrenic nerve could be damaged by the acidic environment The use of local anesthetics has been advocated as a method for reducing postoperative pain local anesthetic intraperitoneal administration has shown good effects on reducing postoperative pain in laparoscopic cholecystectomy and gynecological surgeries . intraperitoneal sodium bicarbonate instillation may neutralize effect of the acid milieu on peritoneal cavity and the phrenic nerve damage which consecutively will lead to a reduction of postoperative pain. Magnesium sulfate, a non-competitive NMDA antagonist, has been proven in animal and human being models to have antinociceptive properties. The antinociceptive effect of magnesium sulfate relieves chronic pain and it can also decrease the duration and intensity of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* age 18:60years
* patients undergoing laparoscopic gynecological surgeries,
* ASA 1&2

Exclusion Criteria:

* patient dissatisfaction for participating in the study
* opioid use within 24 hr before the study
* allergy to the drugs used in the study and alcohol use
* chronic pain syndrome.
* neurological disease.
* steroid treatment

  * conversion of laparoscopic surgery to open surgery
  * use a drain

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gynecological surgeries
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
first rescue analgesia | 24 hour postoperative
  The first request for analgesia will be recorded by the nurse, and in case of pain in VAS more than 3, 1 gm of paracetamol will be administrated as a rescue analgesic if failed fentanyl 100mic will be added

CONTACTS AND LOCATIONS:
Overall Officials: Essam Ezzat Abdel Hakeem, M.D., Study Director — Assiut University